CLINICAL TRIAL: NCT04750941
Title: Pilot Phase II Study of the PI3K Inhibitor Copanlisib in Combination With a Ketogenic Diet in the Treatment of Patients With Relapsed or Refractory Follicular Lymphoma or Endometrial Cancer
Brief Title: Study of Copanlisib and Ketogenic Diet
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: Columbia University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jennifer Amengual, Principal Investigator, Assistant Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS4953
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Follicular Lymphoma; Endometrial Cancer
Keywords: Keto diet; Copanlisib
MeSH Terms: conditions — Lymphoma, Follicular; Endometrial Neoplasms | interventions — copanlisib; Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follicular Lymphoma (FL) (Experimental): The lymphoma study group will enroll 23 patients with FL.
  In cycle 1, patients will first start ketogenic diet for 7 days (Day -6 to Day 0). Only patients who demonstrate compliance and tolerance with the ketogenic diet for all 7 days, as confirmed by pertinent blood and urine tests, will be allowed to continue the study and treatment using copanlisib and the ketogenic diet starting on Day 1. In cycle 2 and beyond, patients will start the ketogenic diet and copanlisib on day 1.
  Interventions: Drug: Copanlisib; Other: Ketogenic Diet
- Endometrial Cancer (EC) (Experimental): The solid tumor group will enroll 19 patients with EC.
  In cycle 1, patients will first start ketogenic diet for 7 days (Day -6 to Day 0). Only patients who demonstrate compliance and tolerance with the ketogenic diet for all 7 days, as confirmed by pertinent blood and urine tests, will be allowed to continue the study and treatment using copanlisib and the ketogenic diet starting on Day 1. In cycle 2 and beyond, patients will start the ketogenic diet and copanlisib on day 1.
  Interventions: Drug: Copanlisib; Other: Ketogenic Diet

INTERVENTIONS:
Drug: Copanlisib — Copanlisib will be infused intravenously on days 1, 8, 15 of each cycle, over 1 hour, of 28-day cycles.
  Other Names: Aliqopa
Other: Ketogenic Diet — In cycle 1, patients will first start the ketogenic diet for 7 days (Day -6 to Day 0).
  Only the patients who demonstrate compliance and tolerance with the ketogenic diet, as confirmed by pertinent blood and urine tests and a diary of diet, will be allowed to continue the study and start copanlisib on Day 1. The ketogenic diet will continue daily throughout the treatment days.
  In cycle 2 and beyond, patients will start the ketogenic diet and copanlisib on day 1.
  The ketogenic diet will then continue daily throughout the treatment days.

SUMMARY:
This is a multicenter, open label, pilot phase II study of the PI3K inhibitor copanlisib in combination with a ketogenic diet in the treatment of patients with one of the following malignancies: (a) relapsed or refractory (R/R) follicular lymphoma (FL), (b) R/R endometrial cancer (EC) with a documented activating mutation in PIK3CA or loss of phosphatase and tensin homolog (PTEN).

DETAILED DESCRIPTION:
As the investigators recently reported ketogenic diet can suppress hyperinsulinemia associated with PI3K inhibitors, leading to potentiation of the anti-tumor effects of PI3K inhibitors. Copanlisib potently inhibits PI3Kα and PI3Kδ. It has been approved for the treatment of relapsed follicular lymphoma, based on ORR of 59% (84 of 142 patients). The CR rate in FL was 14%, and the median progression-free survival was 11.2 months. Copanlisib demonstrated encouraging clinical activity in marginal zone lymphoma (ORR 70% including 9% CR). While these results are clinically meaningful, FL and MZL inevitably develop resistance to copanlisib with time, even in those patients who initially respond to the therapy. Novel strategies to improve the efficacy of copanlisib in FL and MZL, by improving CR and PFS, may transform how to manage these incurable malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* For lymphoma, patients should have measurable disease based on the Lugano Criteria.
* For FL patients must have received at least two lines of prior therapy. There is no upper limit for the number of prior therapies. Tumor tissues of all patients are encouraged to be submitted (optional) prospectively for whole or targeted exome sequencing of key cancer related genes, using the Columbia Combined Cancer Panel (CCCP) or a comparable sequencing platform, such as the MSK-IMPACT 468-gene oncopanel.
* For EC the patients must have recurrent/advanced tumor for which surgical or the systemic curative treatments, or standard therapeutic approaches are not available. The following histologic subtypes are eligible: endometrioid, serous, clear cell, undifferentiated /dedifferentiated, mucinous, squamous, transitional, not-otherwise specified, and mixed celltype.
* Fresh and or archived tumor tissues must be available to (a) establish the diagnosis of the respective malignancies as described in Inclusion Criteria, and (b) be investigated for biomarkers. Patients without historical material or fresh tissue biopsy that is adequate for both diagnosis and correlative studies will not be eligible for the clinical trial.
* Left Ventricular Ejection Fraction (LVEF) > 50%.
* A performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function. All screening labs should be performed within 14 days of treatment initiation.
* HIV positive patients will be eligible as long as the viral load by polymerase chain reaction (PCR) testing is undetectable.
* Female patients of childbearing potential must have a negative pregnancy test within 7 days prior to treatment start.
* Adequate contraception.

Exclusion Criteria:

* The following treatments are prohibited: (a) Chemotherapy (including PI3K inhibitors and other approved or investigational drugs) and monoclonal antibody within 3 weeks; (b) radiotherapy within 2 weeks prior to entering the study; (c) systemic steroids that have not been stabilized (≥ 5 days) to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs.
* Patients that have not recovered from adverse events due to chemotherapy agents administered more than 3 weeks earlier.
* Hypersensitivity to copanlisib or any of its excipients.
* Type I diabetes
* Uncontrolled Type II diabetes mellitus (HbA1c> 7.5%).
* Type II diabetes requiring treatment with a sulfonylurea, meglitinide, or insulin.
* Patients that received major surgery and have not recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients with active, clinically serious infections > CTCAE version 5 Grade 2.
* Patients with known active concurrent malignancy with the following exception: nonmelanoma skin cancer, prostatic intraepithelial neoplasia, or carcinoma in situ of the cervix, prostate cancer that responds to androgen deprivation therapy and has no progression of disease for at least 12 months. If there is a history of prior malignancy, the patient must be disease-free for ≥ 3 years.
* Uncontrolled hypertension, i.e., blood pressure (BP) of ≥ 150/90; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria.
* Concomitant use of strong CYP3A4 inhibitors (defined in the protocol).
* Uncontrolled moderate to severe hypertriglyceridemia (TG>300 mg/dL).
* Myocardial infarction within 6 months of cycle 1, day 1.
* Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV (see Appendix 5).
* An ECG recorded at screening showing evidence of cardiac ischemia.
* Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction < 40% by multigated acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI);
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within 6 months before the start of study medication.
* Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through at least 30 days after the last dose of trial treatment.
* History of nephrolithiasis or nephrolithiasis incidentally discovered during CT screening. *Known selenium deficiency.
* Body mass index (BMI) less than 20.
* An allergy or intolerance to egg, gluten or milk protein.
* History of serious or uncontrolled gout or hyperuricemia.
* Pregnancy, lactation, or breastfeeding.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigators' opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Amengual, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Follicular Lymphoma (FL): In cycle 1, patients with FL will first start the ketogenic diet for 7 days (Day -6 to Day 0). Only patients who demonstrate compliance and tolerance with the ketogenic diet for all 7 days, as confirmed by pertinent blood and urine tests, will be allowed to continue the study and treatment using copanlisib and the ketogenic diet starting on Day 1. In cycle 2 and beyond, patients will start the ketogenic diet and copanlisib on day 1.
- Endometrial Cancer (EC): In cycle 1, patients with EC will first start the ketogenic diet for 7 days (Day -6 to Day 0). Only patients who demonstrate compliance and tolerance with the ketogenic diet for all 7 days, as confirmed by pertinent blood and urine tests, will be allowed to continue the study and treatment using copanlisib and the ketogenic diet starting on Day 1. In cycle 2 and beyond, patients will start the ketogenic diet and copanlisib on day 1.
Period: Overall Study
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were assigned to the EC arm due to enrollment challenges.
Groups:
- Total: Total of all reporting groups
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR will be determined from the number of individuals with a complete response (CR) and number of individuals with a partial response (PR)
Time Frame: Up to 58 weeks or 4 weeks after the last dose
Population: No participants were assigned to the EC arm due to enrollment challenges.
Measure: Number; unit: percent of participants
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
Number analyzed (Participants) | 1 | 0
percent of participants | 100 |

2. Secondary Outcome: Complete Response (CR) Rate
Description: Total number of participants with a CR.
Time Frame: Up to 58 weeks or 4 weeks after the last dose
Population: No participants were assigned to the EC arm due to enrollment challenges.
Measure: Number; unit: percent of participants
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
Number analyzed (Participants) | 1 | 0
percent of participants | 0 |

3. Secondary Outcome: Partial Response (PR) Rate
Description: Total number of participants with a PR.
Time Frame: Up to 58 weeks or 4 weeks after the last dose
Population: No participants were assigned to the EC arm due to enrollment challenges.
Measure: Number; unit: percent of participants
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
Number analyzed (Participants) | 1 | 0
percent of participants | 100 |

4. Secondary Outcome: ORR at the Simon Stage I Analysis
Description: as for outcome 1
Time Frame: Up to 58 weeks or 4 weeks after the last dose
Population: No participants were assigned to the EC arm due to enrollment challenges.
Measure: Number; unit: percent of participants
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
Number analyzed (Participants) | 1 | 0
percent of participants | 100 |

5. Secondary Outcome: Patient Compliance With the Ketogenic Diet
Description: Total # of patients who are compliant with the ketogenic diet.
Time Frame: Up to 58 weeks or 4 weeks after the last dose
Population: No participants were assigned to the EC arm due to enrollment challenges.
Measure: Count of Participants; unit: Participants
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
Number analyzed (Participants) | 1 | 0
Participants | 1 |

ADVERSE EVENTS:
Time Frame: Up to 58 weeks
Description: No participants were assigned to the EC arm due to enrollment challenges.
Arm/Group | Follicular Lymphoma (FL) | Endometrial Cancer (EC)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Follicular Lymphoma (FL) (N=1) | Endometrial Cancer (EC) (N=0)
Weight loss (General disorders) | 1 | 0
Neutrophil count decreased (Immune system disorders) | 1 | 0
Dyspnea (Cardiac disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Bone pain (General disorders) | 1 | 0
Muscle cramp (General disorders) | 1 | 0
Flushing (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT04750941/Prot_SAP_000.pdf